CLINICAL TRIAL: NCT02744261
Title: Evaluating User Perceptions and Experiences of Dual Compartment Microbicide Formulations. Project 5.3: Developing Rectal USPE Measures for Suppositories (Project DRUM-S)
Brief Title: Developing Rectal USPE Measures for Suppositories (Project DRUM-S)
Acronym: DRUM-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: ImQuest Pharmaceuticals, Inc. (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 30048; U19AI101961 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Microbicide Delivery System Perceptibility and Acceptability
Keywords: HIV; STI; Primary Prevention; Topical Microbicides; User Experience; Drug Delivery Systems
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Gels; Green Or

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Formulations (Other): Gel, Suppository 1, Suppository 2
  Interventions: Other: Gel; Other: Suppository 1; Other: Suppository 2

INTERVENTIONS:
Other: Gel — 4 mL
  Other Names: Orange
Other: Suppository 1
  Other Names: Green
Other: Suppository 2
  Other Names: Yellow

SUMMARY:
The purpose of this study is to (a) adapt existing user sensory perception and experience (USPE) items/instruments generated for rectal gel/cream formulations to include USPEs specific to suppository forms for rectal and vaginal use; (b) for both male and female cohorts: to capture the experience of suppository use in the context of receptive anal intercourse (RAI); and (c) for female cohort only: to capture the experience of suppository use in the context of vaginal-penile intercourse (VI), and to compare USPEs of suppository use in the context of RAI to USPEs of suppository use in the context of vaginal-penile intercourse.

DETAILED DESCRIPTION:
HIV prevention is a global public health priority. Providing efficacious prevention methods that have the greatest likelihood of use will have a profound impact on the public's health. Critical to their use is "acceptability." However, current conceptualizations of adherence and acceptability fail to fully articulate and account for patterns of use and non-use. Formulation properties are critically important to both drug delivery and the user experience. Microbicide developers thus have the opportunity to directly control a formulation's impact on acceptability and adherence to product use, as well as biological product performance. Microbicide products can and should be developed such that they achieve performance standards for both these behavioral (user experience) and biological (efficacy) functions. By incorporating the user experience early on in the product development process, developers will have the greatest chance of providing at-risk individuals with the best prevention methods science can provide. Developing prevention products that can be used in the vagina and/or the rectum and that optimize the user experience in both compartments increases the likelihood that these products will be used consistently and correctly. The impact on global public health has the potential to be far-reaching, decreasing HIV and sexually transmitted infections (STI) incidence and prevalence in both women and men.

Methodology and Data Collection: This is a formative mixed methods design in which volunteers (N~20-30; ~10-15 males; ~10-15 females) will first be prescreened for basic study eligibility using a brief questionnaire. Those who are interested in the study and are eligible based on their responses to the prescreen will then complete a STI/HIV screening and pregnancy test (for females).

During the course of the study, participants will evaluate 3 products: 2 distinct suppository formulations and 1 gel formulation that represent a range of rheological and other biophysical properties of potential microbicides being designed for rectal/dual compartment use. Participants will evaluate the experience of suppository use (as compared to gel use) in the context of receptive anal intercourse (RAI) among males and females, and in the context of vaginal intercourse (VI) (females). Each participant will be randomly assigned to the order in which they will evaluate the 3 products. After a sexual encounter that includes RAI/VI and study product use, participants will be required to complete a web survey about their experience with the study product.

ELIGIBILITY:
All participants must meet all of the inclusion criteria to participate in this study.

Inclusion Criteria:

All participants must meet all of the inclusion criteria to participate in this study.

* Eligible male participants must be 18 years of age or older
* Eligible female participants must be 18-45 years of age

Inclusion criteria include men and women who:

* Report receptive anal intercourse (RAI) at least twice in the past 6 months
* Are willing to use each study product in conjunction with RAI on at least one occasion in each data collection period (resulting in a minimum of 3 RAI events during each product evaluation period; on average every 2 weeks, all 3 products across an average of 6 -12 weeks)
* Are willing and able to respond to study data collection systems via phone and internet, attend all study visits, and participate in in-depth qualitative interviews

Additional Inclusion Criteria for Female Volunteers:

* Report vaginal-penile intercourse (VI) at least twice in the past 6 months
* Willing to use each study suppository formulation in conjunction with VI on at least one occasion in each data collection period (resulting in a minimum of 2 vaginal intercourse events during the course of the study)
* Report consistent use of an effective birth control method: e.g., hormonal contraceptive, IUD, bilateral tubal ligation, Essure® or any non-incisional permanent birth control procedure, hysterectomy (partial or total, with/without oophorectomy), partner's vasectomy/salpingectomy

Exclusion Criteria:

* Have a sensitivity or allergy to vaginal, anal, or rectal products
* Have a sensitivity or allergy to any of the ingredients contained in the study products
* Have a sensitivity or allergy to sesame seeds
* Are HIV-positive at baseline, or have a known HIV-positive sexual partner
* Have an active rectal or reproductive tract infection requiring treatment per current CDC guidelines or have other condition that, in the opinion of the investigator/study clinician, make the patient unsuitable for the study or unable to comply with study requirements (Note: HSV seropositivity without active genital lesions is not an exclusion criteria)
* Urinary tract infection (UTI)
* Have current inflammatory bowel disease (IBD) or history of active IBD within last 3 months
* Have any other significant colorectal symptom(s) as determined by medical history, participant self-report, or physical exam (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
* Have any other clinical condition or prior therapy that, in the opinion of the investigator/study clinician, would make the patient unsuitable for the study or unable to comply with the study requirements (including, as determined by medical history, participant self-report, or physical exam: heart disease, high blood pressure, thyroid disease, diabetes, difficulty urinating due to prostate gland enlargement; taking psychotropic medications such as monoamine inhibitors, tricyclic antidepressants, SSRIs)
* Are unwilling to refrain from use of nonoxynol-9 (N9) for the duration of the study
* Are currently enrolled in other rectal or vaginal product studies
* Are unable or unwilling to communicate in English, or
* Are unable or unwilling to give written informed consent

Additional Exclusion Criteria for Female Volunteers:

* Are pregnant or breastfeeding. Pregnancy testing will be conducted at Visits 1-4 (screening and prior to any product use period)
* Have completed menopause (i.e., at least 12 months without menstrual periods)
* Are currently attempting to get pregnant or have an intention to get pregnant during their participation in the study
* Are unwilling to refrain from use of any vaginal product (inclusive of douching; exclusive of tampons during menses) other than study products
* Have clinically significant abnormal pelvic findings and/or findings requiring therapy as a function of clinical exam at Visit 1
* Report being within 30 days of their last pregnancy outcome or gynecologic surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Guthrie, PhD, Principal Investigator — The Miriam Hospital: Centers for Behavioral & Preventive Medicine; Robert Buckheit, PhD, Principal Investigator — ImQuest Pharmaceuticals, Inc.
Locations (1):
- The Miriam Hospital Centers for Behavioral and Preventive Medicine, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
as per individual agreement, provided data safety/confidentiality agreements are met

REFERENCES:
- [Derived] Guthrie KM, Rosen RK, Guillen M, Ramirez JJ, Vargas SE, Fava JL, Ham AS, Katz DF, Cu-Uvin S, Tumilty S, Smith KA, Buckheit KW, Buckheit RW , Jr. Designing Dual Compartment HIV Prevention Products: Women's Sensory Perceptions and Experiences of Suppositories for Rectal and Vaginal Use. AIDS Res Hum Retroviruses. 2022 Jul;38(7):601-610. doi: 10.1089/AID.2021.0038. Epub 2021 Oct 18. PMID 34544269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited (RI, MA USA) via call-lists, flyers, ads, internet/social media, clinics, CBOs, word-of-mouth.
Pre-assignment Details: One female participant was withdrawn prior to use of any study products. She was not able to follow study guidelines and did not use her first study product within the allotted time (I.e., did not use any of the three products).
Groups:
- Females: Female participants that reported user sensory perception experiences for 3 formulations (Orange/Gel, Green/Suppository 1, and Yellow/Suppository 2) during Receptive Anal Intercourse (RAI), and 2 formulations (Green/Suppository 1 and Yellow/Suppository 2) during Receptive Vaginal Intercourse (RVI).
- Males: Male participants that reported user sensory perception experiences for 3 formulations (Orange/Gel, Green/Suppository 1, and Yellow/Suppository 2) during Receptive Anal Intercourse (RAI).
Period: Overall Study
Arm/Group | Females | Males
Started | 17 | 15
Orange/Gel use | 16 | 13
Green/Suppository 1 use | 15 | 15
Yellow/Suppository 2 use | 16 | 15
Completed | 16 (15 pts used all three products (Orange/Gel, Green/Suppository 1, Yellow/Suppository 2); 1 pt used two products (Orange/Gel, Yellow/Suppository 2)) | 15 (13 pts used all three products (Orange/Gel, Green/Suppository 1, Yellow/Suppository 2); 2 pts used two products (Green/Suppository 1, Yellow/Suppository 2))
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Females: Female participants that reported user sensory perception experiences for 3 formulations (Gel, Suppository 1, and Suppository 2) during Receptive Anal Intercourse (RAI), and 2 formulations (Suppository 1 and Suppository 2) during Receptive Vaginal Intercourse (RVI).
- Males: Male participants that reported user sensory perception experiences for 3 formulations (Gel, Suppository 1, and Suppository 2) during Receptive Anal Intercourse (RAI).
- Total: Total of all reporting groups
Arm/Group | Females | Males | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 11 | 4 | 15
  30+ years | 5 | 11 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 0 | 16
  Male | 0 | 15 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1
  White | 10 | 10 | 20
  Asian | 0 | 1 | 1
  American Indian/Alaska Native | 1 | 0 | 1
  More Than One Race (Black/African American, White and American Indian/Alaska Native) | 1 | 0 | 1
  More Than One Race (White and American Indian/Alaska Native) | 0 | 3 | 3
  Other Race (Not specified) | 0 | 1 | 1
  Refused | 3 | 0 | 3
  Hispanic/Latinx | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Yearly Income [Count of Participants; unit: Participants]
  Less than $15,000 | 6 | 0 | 6
  $15,000 - $36,000 | 9 | 3 | 12
  More than $36,000 | 1 | 11 | 12
  Refused to Answer | 0 | 1 | 1
History of STD Diagnosis [Count of Participants; unit: Participants] | 4 | 4 | 8
Vaginal Deliveries [Count of Participants; unit: Participants] — Population: Vaginal deliveries does not apply to Male participants
  Participants
    number analyzed (Participants) | 16 | 0 | 16
    (all) | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: User Perception Scale Scores
Description: USPE Sum of averaged item means/# items (min:max 1:5); 1=Do not agree at all;2=Agree a little;3=Agree somewhat;4=Agree a lot;5=Agree completely
  Products:Gel/Orange, Suppository 1/Green, Suppository 2/Yellow.
  Initial Penetration:Smoothness/lubricity; Initial Lubrication:Coating/lubricating; Spreading Behavior:Ease of stroke, product spread; Product Awareness:Feel during sex (movement, felt betw vaginal/rectal wall-penis); Perceived Wetness:Covering entire vagina/rectum; Stimulating:enhanced pleasure; Messiness:Perceptions of messiness; Leakage:Sensations of leaking during/after sex; Pre-coital Leakage:Product felt/leakage on body or clothes before sex; Naturalness:Sensation of naturalness; leakage looked like vag fluid/cum; Lubricity:Wetness before sex; slipperiness/lubricity during sex; Effortful:Effort needed at penetration; effort difficulty/dryness; Pleasure:Partner's stimulation; Noticeable:messiness, thickness.
  Higher scores=greater agreement re: product characteristics
Time Frame: Web-based survey (same survey; 3 times; one for each formulation) over an average of 6-12 weeks
Population: Numbers analyzed for each scale may differ from overall sample size as a function of sex (and hence opportunity to evaluate) or a non-evaluable scale for a given participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Females | Males
Number analyzed (Participants) | 16 | 15
units on a scale
  SEX: Initial Penetration - RAI (Yellow) | 3.31 (1.14) | 3.36 (1.29)
  SEX: Initial Penetration - RAI (Green): number analyzed (Participants) | 14 | 15
  SEX: Initial Penetration - RAI (Green) | 2.12 (1.45) | 2.62 (1.25)
  SEX: Initial Penetration - RAI (Orange): number analyzed (Participants) | 16 | 12
  SEX: Initial Penetration - RAI (Orange) | 3.06 (1.42) | 3.08 (1.30)
  SEX: Initial Lubrication - RAI (Yellow): number analyzed (Participants) | 15 | 15
  SEX: Initial Lubrication - RAI (Yellow) | 3.63 (1.02) | 3.32 (1.15)
  SEX: Initial Lubrication - RAI (Green): number analyzed (Participants) | 14 | 15
  SEX: Initial Lubrication - RAI (Green) | 2.61 (1.42) | 2.85 (1.17)
  SEX: Initial Lubrication - RAI (Orange): number analyzed (Participants) | 15 | 13
  SEX: Initial Lubrication - RAI (Orange) | 2.84 (1.20) | 3.42 (1.42)
  SEX: Spreading Behavior - RAI (Yellow): number analyzed (Participants) | 15 | 15
  SEX: Spreading Behavior - RAI (Yellow) | 3.44 (1.08) | 3.22 (1.36)
  SEX: Spreading Behavior - RAI (Green): number analyzed (Participants) | 14 | 15
  SEX: Spreading Behavior - RAI (Green) | 2.98 (1.01) | 3.18 (0.88)
  SEX: Spreading Behavior - RAI (Orange): number analyzed (Participants) | 15 | 13
  SEX: Spreading Behavior - RAI (Orange) | 2.98 (1.16) | 3.28 (0.86)
  SEX: Messiness - RAI (Yellow) | 1.98 (0.75) | 1.78 (0.75)
  SEX: Messiness - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Messiness - RAI (Green) | 1.79 (0.67) | 1.82 (0.86)
  SEX: Messiness - RAI (Orange): number analyzed (Participants) | 16 | 13
  SEX: Messiness - RAI (Orange) | 1.77 (0.66) | 1.78 (0.90)
  SEX: Perceived Wetness - RAI (Yellow): number analyzed (Participants) | 13 | 14
  SEX: Perceived Wetness - RAI (Yellow) | 2.77 (0.97) | 2.77 (1.05)
  SEX: Perceived Wetness - RAI (Green): number analyzed (Participants) | 15 | 14
  SEX: Perceived Wetness - RAI (Green) | 2.30 (1.15) | 2.20 (0.67)
  SEX: Perceived Wetness - RAI (Orange): number analyzed (Participants) | 15 | 10
  SEX: Perceived Wetness - RAI (Orange) | 2.43 (1.11) | 2.60 (0.94)
  SEX: Product Awareness - RAI (Yellow): number analyzed (Participants) | 16 | 14
  SEX: Product Awareness - RAI (Yellow) | 2.29 (0.75) | 2.85 (1.11)
  SEX: Product Awareness - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Product Awareness - RAI (Green) | 2.76 (1.10) | 2.63 (0.91)
  SEX: Product Awareness - RAI (Orange): number analyzed (Participants) | 16 | 12
  SEX: Product Awareness - RAI (Orange) | 2.38 (0.82) | 3.32 (0.97)
  SEX: Leakage - RAI (Yellow) | 2.31 (1.01) | 2.17 (0.98)
  SEX: Leakage - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Leakage - RAI (Green) | 1.85 (0.85) | 2.12 (0.87)
  SEX: Leakage - RAI (Orange): number analyzed (Participants) | 16 | 13
  SEX: Leakage - RAI (Orange) | 2.14 (0.93) | 2.29 (0.92)
  SEX: Stimulating - RAI (Yellow): number analyzed (Participants) | 16 | 12
  SEX: Stimulating - RAI (Yellow) | 2.50 (0.95) | 2.93 (1.35)
  SEX: Stimulating - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Stimulating - RAI (Green) | 1.68 (1.09) | 2.43 (1.13)
  SEX: Stimulating - RAI (Orange): number analyzed (Participants) | 16 | 12
  SEX: Stimulating - RAI (Orange) | 2.16 (1.00) | 2.49 (0.94)
  SEX: Naturalness - RAI (Yellow): number analyzed (Participants) | 16 | 13
  SEX: Naturalness - RAI (Yellow) | 2.86 (0.72) | 2.44 (0.59)
  SEX: Naturalness - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Naturalness - RAI (Green) | 1.68 (0.82) | 2.10 (0.67)
  SEX: Naturalness - RAI (Orange): number analyzed (Participants) | 16 | 13
  SEX: Naturalness - RAI (Orange) | 2.31 (0.93) | 2.02 (0.66)
  SEX: Lubricity - RAI (Yellow): number analyzed (Participants) | 16 | 14
  SEX: Lubricity - RAI (Yellow) | 3.25 (1.22) | 2.48 (0.85)
  SEX: Lubricity - RAI (Green): number analyzed (Participants) | 15 | 14
  SEX: Lubricity - RAI (Green) | 2.20 (1.37) | 2.31 (0.91)
  SEX: Lubricity - RAI (Orange): number analyzed (Participants) | 16 | 11
  SEX: Lubricity - RAI (Orange) | 2.54 (1.10) | 2.61 (1.16)
  SEX: Effortful - RAI (Yellow) | 1.75 (0.84) | 1.68 (0.66)
  SEX: Effortful - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Effortful - RAI (Green) | 2.67 (1.37) | 2.12 (1.12)
  SEX: Effortful - RAI (Orange): number analyzed (Participants) | 15 | 13
  SEX: Effortful - RAI (Orange) | 1.80 (0.87) | 1.46 (0.37)
  SEX: Pleasure - RAI (Yellow): number analyzed (Participants) | 15 | 14
  SEX: Pleasure - RAI (Yellow) | 2.78 (1.22) | 3.12 (1.32)
  SEX: Pleasure - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Pleasure - RAI (Green) | 2.04 (1.45) | 2.40 (1.16)
  SEX: Pleasure - RAI (Orange): number analyzed (Participants) | 16 | 12
  SEX: Pleasure - RAI (Orange) | 2.42 (1.45) | 3.06 (1.09)
  SEX: PreCoital Leakage - RAI (Yellow) | 1.35 (0.58) | 1.24 (0.46)
  SEX: PreCoital Leakage - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: PreCoital Leakage - RAI (Green) | 1.18 (0.33) | 1.51 (0.99)
  SEX: PreCoital Leakage - RAI (Orange): number analyzed (Participants) | 16 | 13
  SEX: PreCoital Leakage - RAI (Orange) | 1.21 (0.38) | 1.74 (1.13)
  SEX: Noticeable - RAI (Yellow): number analyzed (Participants) | 16 | 14
  SEX: Noticeable - RAI (Yellow) | 2.27 (1.08) | 2.33 (0.76)
  SEX: Noticeable - RAI (Green): number analyzed (Participants) | 15 | 15
  SEX: Noticeable - RAI (Green) | 2.89 (1.23) | 2.02 (0.70)
  SEX: Noticeable - RAI (Orange): number analyzed (Participants) | 16 | 13
  SEX: Noticeable - RAI (Orange) | 1.96 (0.85) | 2.23 (0.80)
  SEX: Initial Penetration - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Initial Penetration - RVI (Yellow) | 3.73 (0.85) |
  SEX Initial Penetration - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX Initial Penetration - RVI (Green) | 2.44 (1.37) |
  SEX: Initial Lubrication - RVI (Yellow): number analyzed (Participants) | 13 | 0
  SEX: Initial Lubrication - RVI (Yellow) | 3.80 (0.97) |
  SEX: Initial Lubrication - RVI (Green): number analyzed (Participants) | 13 | 0
  SEX: Initial Lubrication - RVI (Green) | 2.89 (1.27) |
  SEX: Spreading Behavior - RVI (Yellow): number analyzed (Participants) | 14 | 0
  SEX: Spreading Behavior - RVI (Yellow) | 3.67 (0.86) |
  SEX: Spreading Behavior - RVI (Orange): number analyzed (Participants) | 14 | 0
  SEX: Spreading Behavior - RVI (Orange) | 3.17 (1.13) |
  SEX: Messiness - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Messiness - RVI (Yellow) | 2.34 (0.79) |
  SEX: Messiness - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Messiness - RVI (Green) | 2.33 (0.86) |
  SEX: Perceived Wetness - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Perceived Wetness - RVI (Yellow) | 3.18 (1.18) |
  SEX: Perceived Wetness - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Perceived Wetness - RVI (Green) | 2.35 (1.13) |
  SEX: Product Awareness - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Product Awareness - RVI (Yellow) | 2.33 (0.78) |
  SEX: Product Awareness - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Product Awareness - RVI (Green) | 2.66 (0.72) |
  SEX: Leakage - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Leakage - RVI (Yellow) | 2.56 (1.04) |
  SEX: Leakage - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Leakage - RVI (Green) | 2.31 (0.97) |
  SEX: Stimulating - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Stimulating - RVI (Yellow) | 2.31 (1.13) |
  SEX: Stimulating - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Stimulating - RVI (Green) | 1.53 (0.91) |
  SEX: Naturalness - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Naturalness - RVI (Yellow) | 2.82 (0.94) |
  SEX: Naturalness - RVI (Green): number analyzed (Participants) | 16 | 0
  SEX: Naturalness - RVI (Green) | 1.88 (1.04) |
  SEX: Lubricity - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Lubricity - RVI (Yellow) | 3.38 (1.02) |
  SEX: Lubricity - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Lubricity - RVI (Green) | 1.91 (1.01) |
  SEX: Effortful - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: Effortful - RVI (Yellow) | 1.23 (0.36) |
  SEX: Effortful - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: Effortful - RVI (Green) | 2.75 (1.60) |
  SEX: Pleasure - RVI (Yellow): number analyzed (Participants) | 14 | 0
  SEX: Pleasure - RVI (Yellow) | 2.55 (1.14) |
  SEX: Pleasure - RVI (Green): number analyzed (Participants) | 14 | 0
  SEX: Pleasure - RVI (Green) | 1.43 (0.77) |
  SEX: PreCoital Leakage - RVI (Yellow): number analyzed (Participants) | 15 | 0
  SEX: PreCoital Leakage - RVI (Yellow) | 1.69 (0.81) |
  SEX: PreCoital Leakage - RVI (Green): number analyzed (Participants) | 15 | 0
  SEX: PreCoital Leakage - RVI (Green) | 1.44 (0.99) |
  SEX: Noticeable - RVI (Yellow): number analyzed (Participants) | 14 | 0
  SEX: Noticeable - RVI (Yellow) | 2.05 (1.05) |
  SEX: Noticeable - RVI (Green): number analyzed (Participants) | 14 | 0
  SEX: Noticeable - RVI (Green) | 3.40 (0.89) |

ADVERSE EVENTS:
Time Frame: 6-12 weeks
Description: Adverse events are separated across arms (Females Gel/Orange, Females Suppository 1/Green, Females Suppository 2/Yellow, Males Gel/Orange, Males Suppository 1/Green, Males Suppository 2/Yellow). Some events are specific to Females and do not apply to Males (Vaginal burning and pain during RVI (receptive vaginal intercourse).
Groups:
- Females Gel/Orange: Female participants that reported user sensory perception experiences for Gel/Orange during Receptive Anal Intercourse (RAI).
- Females Suppository 1/Green: Female participants that reported user sensory perception experiences for Suppository 1/Green during Receptive Anal Intercourse (RAI) and Receptive Vaginal Intercourse (RVI).
- Females Suppository 2/Yellow: Female participants that reported user sensory perception experiences for Suppository 2/Yellow during Receptive Anal Intercourse (RAI) and Receptive Vaginal Intercourse (RVI).
- Males Gel/Orange: Male participants that reported user sensory perception experiences for Gel/Orange during Receptive Anal Intercourse (RAI).
- Males Suppository 1/Green: Male participants that reported user sensory perception experiences for Suppository 1/Green during Receptive Anal Intercourse (RAI).
- Males Suppository 2/Yellow: Male participants that reported user sensory perception experiences for Suppository 2/Yellow during Receptive Anal Intercourse (RAI).
Arm/Group | Females Gel/Orange | Females Suppository 1/Green | Females Suppository 2/Yellow | Males Gel/Orange | Males Suppository 1/Green | Males Suppository 2/Yellow
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/13 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/13 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 2/15 | 2/16 | 2/13 | 1/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Females Gel/Orange (N=16) | Females Suppository 1/Green (N=15) | Females Suppository 2/Yellow (N=16) | Males Gel/Orange (N=13) | Males Suppository 1/Green (N=15) | Males Suppository 2/Yellow (N=15)
Yeast Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The pt mentioned she noticed symptoms of a yeast infection after using the green product for vaginal sex. She experienced vaginal itching and soreness. She had no symptoms about a week after taking an over-the-counter yeast infection suppository.
Vaginal Burning (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Pt experienced vaginal "burning" while having vaginal sex when using green product and it only lasted the remainder of sex, about 4 minutes. She did not experience any symptoms once she was done having vaginal sex.
Anorectal Burning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Female pt experienced burning sensation around anus while partner inserted orange product applicator into her rectum. Male pt experienced a burning sensation inside of rectum 15 seconds after inserting green product and before receptive anal sex.
Pain with RAI Only (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pt experienced pain around her anal opening and inside rectum during receptive anal Intercourse (RAI) while using yellow product. She decided not to continue with sex because it was too painful. Her symptoms resolved once she was done having RAI.
Pain with RAI and RVI (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — While using the yellow product, pt felt discomfort and dryness in her vagina and rectum throughout receptive anal intercourse and receptive vaginal intercourse (two separate days). Her symptoms stopped when she stopped have intercourse.
Burning While Urinating (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pt experienced burning while urinating for 3-4 days during orange/gel product period. Tested positive for gonorrhea. Received an injection and antibiotic pill from his provider. No further treatment needed.
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pt indicated that he typically has a bowel movement after receptive anal intercourse (RAI), but he experienced constipation after RAI while using yellow product. Constipation continued for two days when he was able to have a bowel movement.
Intestinal Cramping/Gassiness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Pt experienced cramping during bowel movement the day after using yellow product during receptive anal intercourse (RAI). Cramping did not persist after bowel movement. Same Pt experienced gassiness the day after using orange product during RAI.

LIMITATIONS AND CAVEATS:
User Sensory Perceptions & Experience (USPE) scales adapted and were used for the first time to evaluate suppository products used by males for receptive anal sex and females for receptive anal sex and receptive vaginal sex.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT02744261/Prot_SAP_000.pdf